CLINICAL TRIAL: NCT06510595
Title: Biomechanical Analysis of Distal Radius (Greenstick) Fracture Healing by Finite Element Method
Brief Title: Biomechanical Analysis of Distal Radius (Greenstick) Fracture Healing
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Hassan Elsheikh, Principal Investigator, University of Huddersfield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005143
Record Dates: First submitted 2024-07-11; First posted 2024-07-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Case-Control study Child A: The child will receive active elbow flexion exercise with electrotherapy.
  Child B: The child will be managed by conservative treatment with brace only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Arm (Experimental): The child will receive active elbow flexion exercise with electrotherapy.
  Interventions: Other: Active Treatment Arm
- Control Treatment Arm (Active Comparator): The child will be managed with conservative treatment using a brace only.
  Interventions: Other: Control Treatment Arm

INTERVENTIONS:
Other: Active Treatment Arm — Electrotherapy:
  Transcutaneous Electrical Nerve Stimulation (TENS) will be placed across the fracture segments. The setting will be adjusted to 2±0.4 Hz sinusoidal wave, with a pulse width set between 50-200 microseconds, and each session will last between 20-30 minutes.
  Active Elbow Flexion Exercise:
  Following the electrotherapy session, the child will perform active assisted elbow flexion exercises with the forearm in a neutral position. This exercise will consist of 3 sets of 15 repetitions to enhance the role of the horizontal components of the brachioradialis muscle force.
  Arms: Active Treatment Arm
Other: Control Treatment Arm — The child will wear a brace as a conservative treatment method.
  Arms: Control Treatment Arm

SUMMARY:
The study will be conducted to investigate the effects of electrical charges (flexoelectric effect) & mechanical brachioradialis muscle bending force on the displacement and strain of fracture gap on children with Distal radius greenstick fracture via finite element method.

DETAILED DESCRIPTION:
Distal radius fractures are common fractures and highly prevalent especially in children, due to skeletal immaturity. They may present as greenstick fractures; due to falling on the outstretched hand during sporting events.

This type of fracture causes deformation and angulation on the cortex layer of bone, while the other side remains intact due to the higher proportion of collagen and flexibility in immature bones, making them more prone to bending rather than breaking completely.

The biomechanical environment plays a dominant role in the process of fracture healing.

It controls the communication network of biological tissues and triggers the complex proliferation process.

This mechanical load is originated from muscle contraction along the axis of bone, which improves the healing process and accelerates the earlier return to weight bearing.

Likewise, the electrical stimulation plays a superior role in acceleration of bone healing. It enhances the cells migration and proliferation process, increases mineralization, and osteogenic genes activation. The bone minerals can generate electromechanical signals through the flexoelectricity effect, which they polarize in response to bending stress force.

While finite element method is an advanced technique and a promising field to simulate the mechanical properties and predict the biomechanical behaviors on the biological structures, no previous research took advantage of both flexoelectricity and mechanical principles to simulate and predict the healing behavior on specific case.

HYPOTHESES:

H0: There will be no significant effect of brachioradialis muscle bending force and flexoelectric effect on strain of distal radius greenstick fracture.

METHODOLOGY

1. The study is analytical and will be conducted by (Finite Element Analysis) study with the following steps:

   * Modelling the radius fracture with angle ≤ 15 degrees.
   * Simulation the strain and displacement of fracture site by computerized mathematical equations with applying brachioradialis muscle force within 10-40 N and electrical charge.
2. Validation the results of computerized simulation by experimental case-control study with the following steps.

Participants :

Child A: The child will receive active elbow flexion exercise with electrotherapy. Child B: The child will be managed by conservative treatment with brace only.

Instrumentation used in treatment:

Transcutaneous Electrical Nerve Stimulation (TENS) is a form of electrotherapy commonly used in physiotherapy to relieve pain. The setting will be adjusted on 2±0.4 Hz sinusoidal wave, pulse width is typically set between 50-200 microseconds and each session lasts between 20-30 minutes.

After the electrotherapy session, active assisted elbow flexion exercise will be applied with forearm in neutral position with 3 × 15 repetition to enhance the role of horizontal components of brachioradialis muscle force.

ELIGIBILITY:
Inclusion Criteria:

* Child with green stick fracture in the distal third of radius bone.
* Child with immobilized brace or splint.
* Angle of fracture is ≤ 15 degrees.

Exclusion criteria:

The participants will be excluded from this study if they have one of the following:

* Other type of bone fracture.
* Osteoporotic bone.
* Neurological diseases.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2024-07-16 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Displacement and strain of fracture gap | Followed up by x-ray weekly for 3:6 weeks.
  The angle of fracture displacement will be measured and followed up by x-ray weekly for 3:6 weeks. A reference line will be determined between proximal and distal points of the radial styloid with the fracture inclination line to identify the radial inclination angle (normal angle 22 -23 degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Enas Youssif, Professor and Chairperson, Study Chair — Musculoskeletal Disorders and its Surgery Faculty of Physical Therapy, Cairo University.; Amr Imam, Professor, Study Director — Applied Mathematics, Damanhour University.; Ahmed Resk Mohammed, Assistant Professor, Study Director — Department of Orthopedic Surgery, Faculty of Medicine, Cairo University; Dina Abd Allah, Lecturer, Study Director — Musculoskeletal Disorders and its Surgery Faculty of Physical Therapy, Cairo University.

REFERENCES:
- [Background] Alierta JA, Perez MA, Garcia-Aznar JM. An interface finite element model can be used to predict healing outcome of bone fractures. J Mech Behav Biomed Mater. 2014 Jan;29:328-38. doi: 10.1016/j.jmbbm.2013.09.023. Epub 2013 Oct 8. PMID 24145150
- [Background] Augat P, Hollensteiner M, von Ruden C. The role of mechanical stimulation in the enhancement of bone healing. Injury. 2021 Jun;52 Suppl 2:S78-S83. doi: 10.1016/j.injury.2020.10.009. Epub 2020 Oct 2. PMID 33041020
- [Background] Bhavsar MB, Han Z, DeCoster T, Leppik L, Costa Oliveira KM, Barker JH. Electrical stimulation-based bone fracture treatment, if it works so well why do not more surgeons use it? Eur J Trauma Emerg Surg. 2020 Apr;46(2):245-264. doi: 10.1007/s00068-019-01127-z. Epub 2019 Apr 6. PMID 30955053
- [Background] Boland MR, Spigelman T, Uhl TL. The function of brachioradialis. J Hand Surg Am. 2008 Dec;33(10):1853-9. doi: 10.1016/j.jhsa.2008.07.019. PMID 19084189
- [Background] Cariati I, Bonanni R, Onorato F, Mastrogregori A, Rossi D, Iundusi R, Gasbarra E, Tancredi V, Tarantino U. Role of Physical Activity in Bone-Muscle Crosstalk: Biological Aspects and Clinical Implications. J Funct Morphol Kinesiol. 2021 Jun 21;6(2):55. doi: 10.3390/jfmk6020055. PMID 34205747
- [Background] Green JS, Williams SC, Finlay D, Harper WM. Distal forearm fractures in children:the role of radiographs during follow up. Injury. 1998 May;29(4):309-12. doi: 10.1016/s0020-1383(97)00208-8. PMID 9743754
- [Background] Gutierrez-Espinoza H, Rubio-Oyarzun D, Olguin-Huerta C, Gutierrez-Monclus R, Pinto-Concha S, Gana-Hervias G. Supervised physical therapy vs home exercise program for patients with distal radius fracture: A single-blind randomized clinical study. J Hand Ther. 2017 Jul-Sep;30(3):242-252. doi: 10.1016/j.jht.2017.02.001. Epub 2017 Mar 22. PMID 28342739
- [Background] Herrmann M, Engelke K, Ebert R, Muller-Deubert S, Rudert M, Ziouti F, Jundt F, Felsenberg D, Jakob F. Interactions between Muscle and Bone-Where Physics Meets Biology. Biomolecules. 2020 Mar 10;10(3):432. doi: 10.3390/biom10030432. PMID 32164381
- [Background] Khare D, Basu B, Dubey AK. Electrical stimulation and piezoelectric biomaterials for bone tissue engineering applications. Biomaterials. 2020 Nov;258:120280. doi: 10.1016/j.biomaterials.2020.120280. Epub 2020 Aug 7. PMID 32810650
- [Background] Kohata K, Itoh S, Takeda S, Kanai M, Yoshioka T, Suzuki H, Yamashita K. Enhancement of fracture healing by electrical stimulation in the comminuted intraarticular fracture of distal radius. Biomed Mater Eng. 2013;23(6):485-93. doi: 10.3233/BME-130774. PMID 24165551
- [Background] Lieber RL, Murray WM, Clark DL, Hentz VR, Friden J. Biomechanical properties of the brachioradialis muscle: Implications for surgical tendon transfer. J Hand Surg Am. 2005 Mar;30(2):273-82. doi: 10.1016/j.jhsa.2004.10.003. PMID 15781349
- [Background] Quadlbauer S, Pezzei C, Jurkowitsch J, Rosenauer R, Kolmayr B, Keuchel T, Simon D, Beer T, Hausner T, Leixnering M. Rehabilitation after distal radius fractures: is there a need for immobilization and physiotherapy? Arch Orthop Trauma Surg. 2020 May;140(5):651-663. doi: 10.1007/s00402-020-03367-w. Epub 2020 Mar 19. PMID 32193679
- [Background] Schmale GA, Mazor S, Mercer LD, Bompadre V. Lack of Benefit of Physical Therapy on Function Following Supracondylar Humeral Fracture: A Randomized Controlled Trial. J Bone Joint Surg Am. 2014 Jun 4;96(11):944-950. doi: 10.2106/JBJS.L.01696. Epub 2014 Jun 4. PMID 24897743